CLINICAL TRIAL: NCT00504673
Title: Comparison of the Effect of Insulin Detemir Versus Insulin NPH Both With Insulin Aspart on Weight Change in Overweight and Obese Subjects With Type 2 Diabetes
Brief Title: Comparison of Insulin Detemir Versus Insulin NPH on Weight Change in Overweight and Obese With Type 2 Diabetes
Acronym: PREDICTIVE™
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN304-1659; 2005-000976-42 (EudraCT Number)
Record Dates: First submitted 2007-07-19; First posted 2007-07-20 (Estimated); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Insulin Detemir; Insulin, Isophane; Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: insulin detemir
Drug: insulin NPH
Drug: insulin aspart

SUMMARY:
This trial is conducted in Europe. The purpose of the trial is to investigate the effect of insulin detemir on weight change in overweight and obese patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* HbA1c: 7.5-11.0%
* BMI: 25-40 kg/m2

Exclusion Criteria:

* Treatment with any OAD (Oral Antidiabetic Drugs) except metformin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 277 (Actual)
Dates: Start 2005-04; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Body weight loss | after 26 weeks of treatment

SECONDARY OUTCOMES:
HbA1c
Incidence of hypoglycaemia

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- A Coruña, Spain

REFERENCES:
- [Derived] Semlitsch T, Engler J, Siebenhofer A, Jeitler K, Berghold A, Horvath K. (Ultra-)long-acting insulin analogues versus NPH insulin (human isophane insulin) for adults with type 2 diabetes mellitus. Cochrane Database Syst Rev. 2020 Nov 9;11(11):CD005613. doi: 10.1002/14651858.CD005613.pub4. PMID 33166419
- [Derived] Fajardo Montanana C, Hernandez Herrero C, Rivas Fernandez M. Less weight gain and hypoglycaemia with once-daily insulin detemir than NPH insulin in intensification of insulin therapy in overweight Type 2 diabetes patients: the PREDICTIVE BMI clinical trial. Diabet Med. 2008 Aug;25(8):916-23. doi: 10.1111/j.1464-5491.2008.02483.x. PMID 18959604
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com